CLINICAL TRIAL: NCT04336150
Title: Effectiveness of Different Hypopressive Exercises for Treating Pelvic Floor Dysfunction in Women: Randomized Controlled Trial
Brief Title: Effectiveness of Different Hypopressive Exercises in Pelvic Floor Dysfunction
Acronym: HIPOSPFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Principal investigator & Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OE13/2017
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Floor Disorders
Keywords: Hypopressive exercises; Pelvic floor muscle trianing; Ultrasound
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypopressive exercisesE (Experimental): Hypopressive exercises described according to Dr. Caufriez
  1. Anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity).
  2. Hypopressive exercises according to the original method described by Dr. Caufriez, which is based on performing the hypopressive maneuver in 33 postures that he described (1,2).
  Interventions: Other: Hypopressive exercises
- Hypopressive exercises&PFM contraction (Experimental): Hypopressive exercises + active pelvic floor muscle contraction:
  1. Anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity).
  2. Hypopressive exercises according to the original method described by Dr.Caufriez, which is based on performing the hypopressive maneuver in 33 postures he described, plus the active contraction of the pelvic floor muscles (PFM) during the hypopressive maneuver.
  Interventions: Other: Hypopressive exercises plus pelvic floor muscle contraction
- Hypopressive maneuver (Experimental): Hypopressive maneuver:
  1. Anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity).
  2. Hypopressive maneuver with transabdominal ultrasound biofeedback.
  Interventions: Other: Hypopressive maneuver
- Hypopressive maneuver&PFM contraction (Experimental): Hypopressive maneuver + pelvic floor muscles contraction:
  1. Anatomical and physiological explanation of the abdomen-pelvic cavity (perineal organs, bone, ligament and muscle structures of the entire abdomen-pelvic cavity).
  2. Hypopressive maneuver plus active contraction of the pelvic floor muscles with transabdominal ultrasound biofeedback.
  Interventions: Other: Hypopressive maneuver plus pelvic floor muscle contraction

INTERVENTIONS:
Other: Hypopressive exercises — See information included in arm/group descriptions.
  Arms: Hypopressive exercisesE
Other: Hypopressive maneuver — See information included in arm/group descriptions.
  Arms: Hypopressive maneuver
Other: Hypopressive exercises plus pelvic floor muscle contraction — See information included in arm/group descriptions.
  Arms: Hypopressive exercises&PFM contraction
Other: Hypopressive maneuver plus pelvic floor muscle contraction — See information included in arm/group descriptions.
  Arms: Hypopressive maneuver&PFM contraction

SUMMARY:
The purpose of the study is to compare the efficacy of different modalities of hypopressive exercises and biofeedback with ultrasound in women with pelvic floor dysfunctions, considering the efficacy of the treatment as improving the specific quality of life related to pelvic floor dysfunctions and improvement of the muscular properties of the pelvic floor muscles.

DETAILED DESCRIPTION:
Female 18-65 years old

Inclusion Criteria:

Women diagnosed with pelvic floor dysfunction by their doctor. With minimum strength of the pelvic floor muscles of 3 according to Modified Oxford Score

Exclusion Criteria:

Women who are pregnant or women who have had a vaginal or caesarean birth in the past six months.

Women whose PFD is severe and the first indication is surgical (POP-Q grade III-IV prolapses).

Women with only urinary incontinence or fecal urgency. Women with pain in the pelvic-perineal region of 3 cm in the visual analog scale, where a score of 0 cm means no pain, and a score of 10cm, the maximum pain that the participant can imagine.

Women who have received pelvic floor physiotherapy treatment in the last 12 months.

Women who are unable to voluntarily contract the pelvic floor muscles, quantified by the Modified Oxford Score by a score less than or equal to 2.

Women with any pathology that may affect the treatment (neurological, gynecological or urological), or with recurrent urinary infection or hematuria.

Women with cognitive limitations to understand the information, answer the questionnaires, consent and / or participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with pelvic floor dysfunction by their doctor.
* With minimum strength of the pelvic floor muscles of 3 according to Modified Oxford Score

Exclusion Criteria:

* Women who are pregnant or women who have had a vaginal or caesarean birth in the past six months.
* Women whose PFD is severe and the first indication is surgical (POP-Q grade III-IV prolapses).
* Women with only urinary incontinence or fecal urgency.
* Women with pain in the pelvic-perineal region of 3 cm in the visual analog scale, where a score of 0 cm means no pain, and a score of 10cm, the maximum pain that the participant can imagine.
* Women who have received pelvic floor physiotherapy treatment in the last 12 months.
* Women who are unable to voluntarily contract the pelvic floor muscles, quantified by the Modified Oxford Score by a score less than or equal to 2.
* Women with any pathology that may affect the treatment (neurological, gynecological or urological), or with recurrent urinary infection or hematuria.
* Women with cognitive limitations to understand the information, answer the questionnaires, consent and / or participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Change in life impact of pelvic floor dysfunction | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be assessed by the PFIQ-7 Spanish version. The PFIQ-7 consists of 3 scales of 7 questions each taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The 3 scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300).
Change in symptoms and quality of life: PFDI-20 | 5 assessments to evaluate change from baseline: at baseline, after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be assessed by PFDI-20 that is both a symptom inventory and a measure of the degree of bother and distress caused by pelvic floor symptoms. The PFDI-20 includes 20 questions and 3 scales. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300 and the higher the score, the worse quality of life. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions collecting data about UI, POP and colorectal and anal symptoms.

SECONDARY OUTCOMES:
Change in pelvic floor muscle strength by manual scale | 5 assessments to evaluate change from baseline after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by Modified Oxford Scale to rate pelvic floor muscle contraction on a scale of 0-5: 0 = no contraction; 1 = minor muscle; 'flicker'; 2 = weak muscle; contraction; 3 = moderate muscle contraction; 4 = good muscle contraction and 5 = strong muscle contraction. T)
Change in pelvic floor muscle strength by dinamometry | 5 assessments to evaluate change from baseline after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by dynamometry (measured in GRAMS).
Change in pelvic floor muscle pasive tone | 5 assessments to evaluate change from baseline after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by dinamometry (measured in GRAMS)
Cahnge in the displacement of the base of the bladder during voluntary contraction of the pelvic floor | 5 assessments to evaluate change from baseline after the intervention period (2 months from baseline), 3 months, 6 months and 12 months after the intervention.
  It will be measured by Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: María Torres-Lacomba, PhD, Principal Investigator — University of Alcalá
Locations (1):
- María, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No